CLINICAL TRIAL: NCT01537406
Title: Long Term Outcomes of A Multicentre Controlled Clinical Trial of Breast Irradiation Using Intensity-Modulated Radiation Therapy
Brief Title: Long Term Outcomes of Breast Intensity-Modulated Radiation Therapy
Acronym: BIMRT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: BCCABreastIMRT
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: BREAST IRRADIATION USING INTENSITY MODULATED RADIATION THERAPY
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: BREAST IRRADIATION USING INTENSITY-MODULATED RADIATION THERAPY — LONG TERM OUTCOMES OF A MULTICENTRE CONTROLLED CLINICAL TRIAL OF BREAST IRRADIATION USING INTENSITY-MODULATED RADIATION THERAPY

SUMMARY:
The purpose of this study is to evaluate the frequency of chronic breast pain about 8 years after the delivery of the radiation treatment, and to compare the frequency between subjects that received breast Intensity-Modulated Radiation Therapy (IMRT) and those that received standard wedge radiotherapy. The cosmetic result, meaning how similar is the treated breast compared to the non-treated breast, will be assessed. Also, the occurrence of delayed radiation treatment side effects including tiny red vessels in the skin, breast indurations (hardening of the skin), skin discoloration, oedema (swelling of the breast), and skin dryness will be captured.

DETAILED DESCRIPTION:
The Canadian breast IMRT clinical trial accrued 358 subjects between July 2003 to March 2005. Those subjects were randomised between standard radiotherapy using 2D wedge compensation and breast IMRT. Subjects were treated in Toronto, Ontario, or in Victoria, British Columbia. Subjects and assessors were carefully blinded to the treatment arm. The clinical trial was funded by the Canadian Institute for Health Research (CIHR) and one of the four objectives of the application was to "To record late skin toxicity occurrence, fibrosis and telangiectasia, in women receiving breast IMRT and conventional irradiation technique".

The investigators are proposing to invite women who participated in the trial to return to their treatment centre during 2011-2013 for a follow-up assessment at eight years after randomisation to record relevant long-term outcomes including the effect of improved homogeneity with IMRT on the occurrence of late radiation therapy side-effects cosmetic outcome and Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* Subject randomised in the initial breast IMRT randomized trial will be eligible for this new study

Exclusion Criteria:

* Subjects who have experienced a recurrence (invasive or in situ) in the breast will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer subjects treated in Toronto, Ontario, or in Victoria, British Columbia that participated in The Canadian breast IMRT clinical trial between July 2003 to March 2005.
Sampling Method: Probability Sample
Enrollment: 314 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Does breast IMRT reduces the occurrence of chronic breast pain after radiation therapy. | 8 years post RT
  A Self pain measurement questionnaire using Visual analog scale (VAS) The nurse coordinator will assess the subject's breast pain due to radiation using the CTCAE 4.0 scale Subjects will complete a Self pain measurement short form of the McGill pain questionnaire

SECONDARY OUTCOMES:
Does breast IMRT reduce the occurrence of late radiation therapy side effects | 8 years post RT
  A EORTC Breast Cancer Rating System for the cosmetic assessment RTOG/EORTC Late Radiation Morbidity Scoring Scheme Cosmetic outcome of the treated breast as compared with the untreated using the Harvard criteria Digital images (photographs) will be taken of the treated and untreated breasts.
  Breast Cancer Treatment Outcome Scale (BCTOS) questionnaire
Does breast IMRT effect long term QOL | 8 Years post RT
  A EORTC Breast Cancer Rating System for the cosmetic assessment RTOG/EORTC Late Radiation Morbidity Scoring Scheme Cosmetic outcome of the treated breast as compared with the untreated using the Harvard criteria Digital images (photographs) will be taken of the treated and untreated breasts.
  Breast Cancer Treatment Outcome Scale (BCTOS) questionnaire
Does IMRT effect local recurrence rates, overall and disease free survivals. | 8 years post RT
  Data collection of local recurrences, overall and disease free survivals.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Pignol, MD, Principal Investigator — Odette Cancer Centre; Pauline Truong, MD, Principal Investigator — BCCA - Vancouver Island Cancer Centre; Ivo Olivotto, MD, Principal Investigator — BCCA - Vancouver Island Cancer Centre
Locations (2):
- Canada (2):
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - Odette Cancer Centre, Toronto, Ontario